CLINICAL TRIAL: NCT04889573
Title: Immunoglobulin Gene Rearrangement and Repair in Healthy Donors
Acronym: R2IGH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 87RI20_0074 (R2IGH)
Record Dates: First submitted 2021-05-05; First posted 2021-05-17 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteers
Keywords: B-cells; BCR; VDJ rearrangement; SHM; CSR; LSR; Ig; HTS; normal values
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Blood sample (Experimental)
  Interventions: Genetic: Blood sample

INTERVENTIONS:
Genetic: Blood sample — The blood samples will be collected from healthy volunteers : 7 tubes of 7 ml with anti-coagulant Héparine Lithium and 1 tube of 7ml with anti-coagulant EDTA

SUMMARY:
B-cells ensure humoral immune response against antigens (Ag) thanks to their receptor (BCR). V(D)J rearrangement, somatic hypermutation, immunoglobulin (Ig) class switch and locus suicide recombination are mutational/recombinational processes targeting Ig loci influencing BCR expression. Study of these events is essential for B cell function analysis. Our project will provide the normal reference values using high throughput sequencing-based protocols.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers aged between 18 and 70
* volunteers free from lymphoid hemopathy, immune deficiency and autoimmune disease.

  3 categories : volunteers between 18 and 34 years of age, volunteers between 35 and 50 years of age, volunteers between 51 and 69 years of age.

Exclusion Criteria:

* any recent vaccination (< 4 weeks)
* tumoral pathology
* lymphoïd hemopathy
* immune deficiency
* autoimmune disease
* transplanted patients
* inflammatory / systemic diseases
* hypersensitivity or allergies
* treatments likely to modify the immune response :

  * calcineurin inhibitors: ciclosporin, tacrolimus -antimetabolite: azathioprine, mycophenolate mofetil / mycophenolic acid, 6-mercaptopurine, methotrexate
  * cyclophosphamide
  * antilymphocyte serum (rabbit, horse)
  * mTOR inhibitors: everolimus, sirolimus
  * anti-CD25 (anti IL2-R): basiliximab, dacliximab -belatacept (anti CD80-86)
  * abatacept (CTLA4-Ig)
  * OKT3 (Muronomab-CD3, anti-CD23)
  * glucocorticoids: methylprednisolone, prednisone, prednisolone.
  * entuzumab (anti-CD52)
  * rituximab, ocrelizumab (anti-CD20)
  * eculizumab (anti-C5)
  * anakinra (analogue IL1-RA)
  * leflunomide (dihydroorotate dehydrogenase inhibition)
  * bortezomib (proteasome inhibitor)
  * fingolimod (S1P receptor antagonist)
  * alentuzumab (anti CD52)
  * Ig G -antiTNF (etanercept, infliximab, adalimumab, certolizumab)
  * vedolizumab (Anti-integrin α4β7 Ab)
  * ustekinumab (anti-IL12)
  * natalizumab (anti-integrin a4)
  * mitoxantrone (topoisomerase type II inhibitor)
  * tocilizumab (anti-IL6)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Frequency of use of the V, D and J genes in VDJ rearrangements | through study completion, an average of 18 months

SECONDARY OUTCOMES:
Percentage of HyperMutation Somatic (SHM) in VDJ regions | through study completion, an average of 18 months
Nature of HyperMutation Somatic (SHM) | through study completion, an average of 18 months
  transitions and transversions
Ig class switching (CSR) and recombination suicide of the IgH locus (LSR) junctions | through study completion, an average of 18 months
  number of CSR and LSR junctions
Frequency of g class switching (CSR) and recombination suicide of the IgH locus (LSR) junctions | through study completion, an average of 18 months
  frequency of CSR and LSR junctions according to their structure

CONTACTS AND LOCATIONS:
Locations (1):
- Limoges University Hospital, Limoges, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al Jamal I, Parquet M, Guiyedi K, Aoufouchi S, Le Guillou M, Rizzo D, Pollet J, Dupont M, Boulin M, Faumont N, Boutouil H, Jardin F, Ruminy P, El Hamel C, Lerat J, Al Hamaoui S, Makdissy N, Feuillard J, Gachard N, Peron S. IGH 3'RR recombination uncovers a non-germinal center imprint and c-MYC-dependent IGH rearrangement in unmutated chronic lymphocytic leukemia. Haematologica. 2024 Feb 1;109(2):466-478. doi: 10.3324/haematol.2023.282897. PMID 37496419